CLINICAL TRIAL: NCT06071897
Title: Introduction of Induction Chemoimmunotherapy Regimen for the Treatment of Pediatric Patients With Stage 4 High-risk Neuroblastoma and Ganglioneuroblastoma Older 18 Months
Brief Title: Induction Chemoimmunotherapy for Patients With High-risk Neuroblastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI-2023-08
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Neuroblastoma; Ganglioneuroblastoma
MeSH Terms: conditions — Neuroblastoma; Ganglioneuroblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental): * days of 21 days schedule N5
  * Vincristine 1,5 mg/m2 i.v., day 1*
  * Etoposide 100 mg/m2 i.v. , days 1-4*
  * Cisplatin 100 mg/m2 i.v., days 1-4* N6
  * Vincristine 1,5 mg/m2 i.v. on days 1, 8*
  * Dacarbasine 200 mg/m2 i.v., days 1-5*
  * Ifosphamide 1500 mg/m2 i.v, days 1-5*
  * Doxorubicin 30 mg/m2 i.v, days 6, 7*
  N5Q
  * N5 (see above)
  * Dinutuximab beta 10 mg/m2 i.v., days 5-9*
  G-CSF (granulocyte colony-stimulating factor) 5 mcg/kg s.c. on day 9 until the ANC is more than 2000 /ml or until counts have recovered for the next cycle of therapy
  N6Q
  * N6 (see above)
  * Dinutuximab beta 10 mg/m2 i.v., days 6-10*
  G-CSF (granulocyte colony- stimulating factor) 5 mcg/kg s.c. on day 10 until the ANC is more than 2000 /ml or until counts have recovered for the next cycle of therapy
  Delayed surgery (if needed) will be done after the 4th or 6th course of induction therapy and stem cells apheresis after the 2nd-5th course of induction therapy.
  Interventions: Drug: monoclonal antibodies GD2

INTERVENTIONS:
Drug: monoclonal antibodies GD2 — Main target of this trial is to estimate tolerability and toxicity of combination of standard chemotherapy (N5 and N6) with anti-GD2 MAB
  N5Q. N5 (see above) Dinutuximab beta 10 mg/m2 i.v., days 5-9*
  N6Q. N6 (see above) Dinutuximab beta 10 mg/m2 i.v., days 6-10*
  G-CSF (granulocyte colony-stimulating factor) 5 mcg/kg s.c. on day 9 until the ANC is more than 2000 /ml or until counts have recovered for the next cycle of therapy

SUMMARY:
The modern strategy of therapy of high-risk neuroblastoma, stage 4, consists of three phases - induction, consolidation and post- consolidation. Still current approaches demonstrates insufficient levels of ORR (overall response rate), OS (overall survival) and EFS (event free survival).

NB-HR-2023 (neuroblastoma high risk) protocol aimed to investigate tolerability and toxicity and potential improvement of ORR, OS and EFS by overcoming of tumor heterogeneous drug resistance using the synergistic interaction of cytostatic and immunobiological agents in the induction. Protocol include the combination of standard chemotherapy (N5 and N6) with anti-GD2 MAB, which is potentially expected to improve outcomes in patients with high-risk neuroblastoma and ganglioneuroblastoma, 4th stage older 18 months.

Currently, treatment with combinations of cytostatics with immunobiological agents is limited due to the risk of complications, which, nevertheless, is controlled with proper monitoring and concomitant therapy. Still no data about use of combination of standard chemotherapy (N5 and N6) with ch14.18/CHO MAB (dinutuximab beta) in induction in primary patients with neuroblastoma.

Prospective, interventional trial include patients with neuroblastoma and ganglioneuroblastoma, 4th stage of the high-risk group older 18 months, who will receive combination of standard induction chemotherapy (N5 and N6) with anti-GD2 MAB. Consolidation and post consolidation chemotherapy courses are not the subjects for analysis.

Patients with high-risk neuroblastoma and ganglioneuroblastoma, stage 4, older 18 months who receive combination of standard induction chemotherapy (N5 and N6) with anti-GD2 MAB at the Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology Delayed surgery (if needed) will be done after the 4th or 6th course of induction therapy and stem cells apheresis after the 2nd-5th course of induction therapy.

DETAILED DESCRIPTION:
The modern strategy of therapy of high-risk neuroblastoma, stage 4, consists of three phases - induction, consolidation and post- consolidation. Still current approaches demonstrates insufficient levels of ORR (overall response rate), OS (overall survival) and EFS (event free survival). NB-HR-2023 protocol aimed to investigate potential improvement of ORR, OS and EFS by overcoming of tumor heterogeneous drug resistance using the synergistic interaction of cytostatic and immunobiological agents in the induction. Protocol include the combination of standard chemotherapy (N5 and N6) with anti-GD2 MAB, which is potentially expected to improve outcomes.

Currently, treatment with combinations of cytostatics with immunobiological agents is limited due to the risk of complications, which, nevertheless, is controlled with proper monitoring and concomitant therapy. Still no data about use of combination of standard chemotherapy (N5 and N6) with anti-GD2 MAB in induction.

Main target of this trial is to estimate tolerability and toxicity of combination of standard chemotherapy (N5 and N6) with anti-GD2 MAB Prospective, interventional trial include patients with high-risk neuroblastoma and ganglioneuroblastoma, 4th stage older 18 months, who will receive combination of standard induction chemotherapy (N5 and N6) with anti-GD2 MAB. Consolidation and post-consolidation chemotherapy courses are not the subjects for analysis.

Patients (n=15) with high-risk neuroblastoma and ganglioneuroblastoma, 4th stage , who receive combination of standard induction chemotherapy (N5 and N6) with anti-GD2 MAB at the Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology.

Patients to be enrolled should met the eligibility criteria (see below) and will receive the induction therapy: two courses of standard chemotherapy and four courses of combination of anti-GD2 МАB ch14.18/CHO (dinutuximab beta).

N5Q cycle: cisplatin (40 mg/m2 per day, IV, in days 1-4) + etoposide (100 mg/m2 per day, IV, days 1-4) + vincristine (1,5 mg/m2 per day, IV, day 1 + dinutuximab beta (10 mg/m2 per day, IV, Days 5-9) N6Q cycle: vincristine (1.5 mg/m2 per day, IV, days 1, 8) + dacarbazine (200 mg/m2 per day, IV, days 1-5) + ifosfamide (1500 mg/m2 per day, IV, days 1-5) + doxorubicin (30 mg/m2 per day, IV, days 6, 7) + dinutuximab beta (10 mg/m2 per day, IV days 6-10).

Delayed surgery (if needed) will be done after the 4th or 6th course of induction therapy and stem cells apheresis after the 2nd-5th course of induction therapy.

Interim analyses will be carried out in 1, 2 and 3 years from the first patient enrollement.

The final analysis with the assessment of the ORR, OS, EFS of patients will be carried out in 1 year and 3 years from the date of inclusion of the last patient in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Verified diagnosis of neuroblastoma or ganglioneuroblastoma (ICD-10 codes C47.3, C47.4, C47.5, C47.6, C47.8, C47.9, C48, C74.1, C74.9, C76.0, C76.1, C76.2, C76.7, C76.8).
* High-risk patients in accordance with the risk stratification of to the GPOH-NB2004 protocol with stage 4 according to the International Neuroblastoma Staging System (INSS) from 18 months of life to 18 years.
* ≥ 70% estimation by Lansky or Karnowski scale at the at the start point of chemoimmunotherapy.
* Life expectancy ≥ 12 weeks from therapy initiation
* No signs of drug-induced neuropathy or neuropathic pain.
* Adequate liver function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) activity < 5 values of the upper limit of the norm (VGN).
* Adequate renal function: creatinine clearance or glomerular filtration rate (GFR) > 60 ml/min/1.73 m2.
* Coagulogram parameters: prothrombin index (PTI) 70-120%, activated partial thromboplastin time (APTT) < 36 s.
* Absence of clinical signs of heart failure, left ventricular ejection fraction (LVEF) ≥ 55%.
* Assessment of the function of the respiratory system (saturation on the pulse oximeter > 94% without the use of oxygen, there is no respiratory disturbance at rest), the absence of pathology during chest X-ray.

Exclusion Criteria:

* Neuroblastoma or ganglioneuroblastoma of the low-risk group or intermediate-risk group, by NB 2004 protocol and disease staging according to INSS (stages 1-3 and 4s without apmplification of MYCN gene, stage 4 in patients under 18 months of age) and high-risk patients with stages 1-3/4s with amplification of MYCN gene.
* Presence in anamnesis of acute intolerance reactions or contraindications to the main chemotherapeutic, immunobiological agents and any concomitant therapy drugs used within the framework of this clinical trial protocol.
* Pregnancy due to the high teratogenic activity and toxicity of drugs used in the clinical trial protocol. A pregnancy test is indicated for patients of childbearing age.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the Tolerability of the induction chemoimmunotherapy regimen based of courses N5 and N6 with anti-GD2 MAB measured by number of AEs (grade 1-2-3-4-5 measured by CTCAE v.5.0) | 3 years after the start of therapy
Estimate the toxicity of the induction chemoimmunotherapy regimen based of courses N5 and N6 with anti-GD2 MAB measured by number of AEs (grade 1-2-3-4-5 measured by CTCAE v.5.0) | 3 years after the start of therapy

SECONDARY OUTCOMES:
ORR | At the end of cycle 6 (each cycle is 21 days)
  To assess the overall response rate (ORR, %) in patients received the induction combination of standart chemotherapy (N5) with anti-GD2 MAB
ORR | At the end of cycle 6 (each cycle is 21 days)
  To assess the overall response rate (ORR, %) in patients received the induction combination of standart chemotherapy (N6) with anti-GD2 MAB
OS | 1 and 3 years after completetion of 6th course of induction ( each cycle is 21 days)
  To assess overall survival (OS, %) after combination of standart chemoimmunotherapy (N5 and N6) with anti-GD2 MAB
EFS | 1 and 3 years after completetion of 6th course of induction ( each cycle is 21 days)
  To assess event free survival (EFS, %) after combination of standart chemoimmunotherapy (N5 and N6) with anti-GD2 MAB

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No